CLINICAL TRIAL: NCT06195826
Title: Gravity Versus Pump Infusion of Distending Media for Hysteroscopic Myomectomy: A Retrospective Cohort Study
Brief Title: Gravity Versus Pump Infusion of Distending Media for Hysteroscopic Myomectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 112180-E
Record Dates: First submitted 2023-12-05; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Hysteroscopic Myomectomy
MeSH Terms: interventions — Infusion Pumps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- gravity infusion: women who received hysteroscopic myomectomy with gravity infusion method
  Interventions: Procedure: Gravity infusion
- pump infusion: women who received hysteroscopic myomectomy with pump infusion method
  Interventions: Procedure: Pump infusion

INTERVENTIONS:
Procedure: Gravity infusion — hysteroscopic myomectomy with the gravity infusion method
  Groups: gravity infusion
Procedure: Pump infusion — hysteroscopic myomectomy with the pump infusion method
  Groups: pump infusion

SUMMARY:
To compare the perioperative outcome between the gravity versus pump infusion groups in women who received hysteroscopic myomectomy

ELIGIBILITY:
Inclusion Criteria:

* >20 years old women
* women who received hysteroscopic myomectomy

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with uterine myoma
Study Population: Patients who received hysteroscopic myomectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Infusion volume of distension medium | 1 week
  Infusion volume (mL) of distension medium in the uterine cavity between the gravity and pump infusion methods for hysterosopic myomectomy

SECONDARY OUTCOMES:
Intraoperative blood loss | 1 week
  Intraoperative blood loss (mL) between the gravity and pump infusion methods for hysterosopic myomectomy
Postoperative pain | 1 week
  Postoperative pain (visual analogue scale 0-10) in the recovery room between the gravity versus pump infusion methods for hysterosopic myomectomy.
Surgical time | 1 week
  Surgical time (minutes) between the gravity versus pump infusion methods for hysterosopic myomectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan